CLINICAL TRIAL: NCT00504894
Title: Neuroimaging the Effects of Intravenous Anesthetic on Amygdala Dependent Memory Processes
Acronym: Amygdala
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: One study drug (thiopental) became commercially unavailable
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0701008933; K08GM083213 (NIH)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: N/A healthy volunteers
MeSH Terms: interventions — Propofol; Thiopental

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo given in low dose to gauge subject's responses to visual stimuli.
  Interventions: Drug: Placebo
- Propofol (Active Comparator): Propofol given at 0.90 μgml-1 to gauge subject's responses to visual stimuli.
  Interventions: Drug: Propofol
- Thiopental (Active Comparator): Thiopental given at 3.0 μgml-1 to gauge subject's responses to visual stimuli.
  Interventions: Drug: Thiopental

INTERVENTIONS:
Drug: Placebo — A low dose given intravenously one time for just under an hour while the subject is shown visually stimulating images in an MRI machine.
  Arms: Placebo
Drug: Propofol — A low dose of propofol 0.90 μgml-1, given intravenously while the subject is shown visually stimulating images in an MRI machine.
  Arms: Propofol
Drug: Thiopental — A low dose of thiopental 3.0 μgml-1, given intravenously while the subject is shown visually stimulating images in an MRI machine.
  Arms: Thiopental

SUMMARY:
This study involves 60 healthy volunteers aged between 18 and 50 recruited from the general community. It involves doing a set of simple memory tests while inside a fMRI machine. The subject is given a very low dose of an anesthetic drug intravenously while in the scanner. The subject then sees a sequence of pictures on a screen, and presses a button if they remember seeing the picture before. While this is happening, the scanner will be capturing images that tell us what parts of the brain are active. Hypothesis: patterns of hippocampal and amygdala activation during the encoding and retrieval of memory,as measured by fMRI, will be altered by intravenous anesthetics such that suppression of hippocampal and amygdala activities will be dissociable. This dissociation pattern will be different between the drugs propofol and thiopental.

DETAILED DESCRIPTION:
Background: Subclinical doses of propofol produce anterograde amnesia, characterized by an early failure of memory consolidation. It is unknown how propofol affects the amygdala-dependent emotional memory system, which modulates consolidation in the hippocampus in response to emotional arousal and neurohumoral stress. We present an event-related functional magnetic resonance imaging study of the effects of propofol on the emotional memory system in human subjects.

Methods: Sixty healthy subjects were randomized to receive propofol, at an estimated brain concentration of 0.90 μgml-1, thiopental, at an estimated brain concentration of 3.0 μgml-1, or placebo. During drug infusion, emotionally arousing and neutral images were presented in a continuous recognition task, while blood-oxygen-level-dependent activation responses were acquired. After a drug-free interval of 2 h, subsequent memory for successfully encoded items was assessed. Imaging analysis was performed using statistical parametric mapping and behavioural analysis using signal detection models.

ELIGIBILITY:
Inclusion Criteria:

* age b/w 18 and 50
* right-handed
* minimum of high school education
* fluent in English
* normal vocabulary

Exclusion Criteria:

* any significant medical/psychiatric comorbidity
* deficit in vision or hearing that would impede the study
* allergies to any of the study drugs, to soybeans, or eggs.
* history of head trauma
* family history of major psychiatric illness
* body mass index > 30 kg/m2
* claustrophobia
* prior exposure to IAPS pictures
* pregnancy
* permanent metal objects anywhere in the body
* a personal/family history of any porphyria

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kane Pryor, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pryor KO, Root JC, Mehta M, Stern E, Pan H, Veselis RA, Silbersweig DA. Effect of propofol on the medial temporal lobe emotional memory system: a functional magnetic resonance imaging study in human subjects. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i104-i113. doi: 10.1093/bja/aev038. PMID 26174294

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol: Propofol give at 0.90 μgml-1 to gauge subject's responses to visual stimuli.
  Propofol: A low dose of propofol 0.90 μgml-1, given intravenously while the subject is shown visually stimulating images in an MRI machine.
- Thiopental: Thiopental give at 3.0 μgml-1 to gauge subject's responses to visual stimuli.
  Thiopental: A low dose of thiopental 3.0 μgml-1, given intravenously while the subject is shown visually stimulating images in an MRI machine.
Period: Overall Study
Arm/Group | Placebo | Propofol | Thiopental
Started | 20 | 21 | 19
Completed | 17 | 18 | 19
Not Completed | 3 | 3 | 0
Not completed — fMRI technical problems | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Infusion technical problems | 0 | 1 | 0
Not completed — poor subject data | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Propofol | Thiopental | Total
Number analyzed (Participants) | 20 | 21 | 19 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 29] | 25 [23 to 26] | 24 [22 to 32.5] | 25 [22 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 13 | 42
  Male | 5 | 7 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Blood-oxygen-level-dependent Significant Activation Cluster
Description: Three anatomical regions for which there was an a priori mechanistic hypothesis were assessed using standard small volume correction: (i) the amygdala, bilaterally; (ii) the hippocampus, bilaterally; and (iii) the parahippocampus, bilaterally. Using single-tailed t tests, a priori regions were reported as significant if the initial uncorrected voxel-wise P value was < 0.001, and then the P value was < 0.05 after family-wise error correction for multiple comparisons in the hypothesized anatomical region. For non-hypothesized regions outside the medial temporal lobe, findings were reported as significant if the initial uncorrected voxel-wise P value was < 0.001, and then the P value was < 0.05 after family-wise error correction for multiple comparisons across the whole brain. Clusters containing voxel maxima at these thresholds are reported.
Time Frame: for 90 minutes after the drug/placebo was commenced
Population: Of the 20 placebo subjects recruited, 3 subjects' data was excluded due to technical problems or poor quality.
  Of the 21 propofol subjects recruited, 3 subjects' data was excluded due to technical problems, poor quality, or subject withdrawal.
  Of the 19 thiopental subjects recruited, no subjects' data was excluded.
Measure: Number; unit: BOLD significantly activated clusters
Arm/Group | Placebo | Propofol | Thiopental
Number analyzed (Participants) | 17 | 18 | 19
BOLD significantly activated clusters
  Right Amygdala | 1 | 1 | 1
  Left Amygdala | 1 | 1 | 1
  Right Hippocampus | 1 | 0 | 0
  Left Hippocampus | 1 | 0 | 1
  Right Parahippocampal Cortex | 0 | 0 | 0
  Left Parahippocampal Cortex | 0 | 0 | 0

2. Secondary Outcome: Blood-oxygen-level-dependent Significant Activation Cluster for Positive Sequential Memory
Description: as for outcome 1
Time Frame: for 90 minutes after the drug/placebo was commenced
Population: as for outcome 1
Measure: Number; unit: BOLD significantly activated clusters
Arm/Group | Placebo | Propofol | Thiopental
Number analyzed (Participants) | 17 | 18 | 19
BOLD significantly activated clusters
  Right Amygdala | 0 | 0 | 0
  Left Amygdala | 1 | 0 | 0
  Right Hippocampus | 0 | 0 | 1
  Left Hippocampus | 1 | 0 | 0
  Right Parahippocampal Cortex | 0 | 0 | 0
  Left Parahippocampal Cortex | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Propofol | Thiopental
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No